CLINICAL TRIAL: NCT05044247
Title: The Effect of Both Ultrasound and Fluoroscopy Guide Erector Spinae Plane Blocks in Patient Undergo Breast Surgery or Pain Intervention Procedures
Brief Title: The Effect of Both Ultrasound and Fluoroscopy Guide Erector Spinae Plane Blocks
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202008018RINC
Record Dates: First submitted 2021-09-05; First posted 2021-09-14 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2020-09

CONDITIONS: Pain, Chronic; Pain, Postoperative
MeSH Terms: conditions — Chronic Pain; Pain, Postoperative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ESP block (Experimental): ESP block under mixed local anesthetics, betamethasone agent
  Interventions: Procedure: ESP blocks

INTERVENTIONS:
Procedure: ESP blocks — ultrasound and fluoroscopy to identify the spread of drug

SUMMARY:
Since the original publication on the erector spinae plane (ESP) block in 2016, the technique of the ESP block has evolved significantly in the last few years. Current reports suggest that the ESP block provides adequate analgesia in thoracic and abdominal sites in a post-surgical and chronic pain patient. However, there were still inconsistencies and unclear spread of local anesthetics in ultrasound guide ESP block.

This study focusing on the spread of local anesthetic in ESP block under ultrasound and fluoroscopy and possible mechanisms of action.

DETAILED DESCRIPTION:
The erector spinae plane (ESP) block was first described by Forero et al. Considering the spread of local anesthetic in the ESP block, it can block more extensive spinal nerves. Therefore, since the first publication, the ESP block has been reported as an effective analgesic for several types of pain and has been used mainly in thoracic surgery. It also used in abdominal surgery, nephrectomy, hernia surgery, and hip surgery, among others. Additionally, the ESP block used not only acute pain management but also chronic pain management.

The spread of local anesthetic in the ESP block investigated in several ways, such as computed tomography (CT) imaging of cadavers, fluoroscopy, chest radiography, and patients' CT imaging. These investigations show that local anesthetics in the ESP block spread to the upper and lower sides of the interfascial plane between the erector spine muscle and the underlying transverse process. Additionally, the local anesthetic spreads beyond the transverse process to reach the costotransverse junctions, after which it permeates the paravertebral space.

Despite the many publications on ESP blocks, there are still inconsistencies and unclear aspects of the technique, such as the spread of local anesthetic and action mechanisms This study focuses on the spread of local anesthetic in ESP block under ultrasound and fluoroscopy and possible mechanisms of action.

ELIGIBILITY:
Inclusion Criteria:

1. Thirty-five patients in each group of breast tumor surgery and pain intervention procedure patients.
2. Age > 20

Exclusion Criteria:

1. Unable to complete questionnaires.
2. With coagulopathy
3. History of thoracic spine trauma or surgery.
4. Allergy to contrast local anesthetics and medium (Iohexol)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Pain scale | 12 months
  reduction of Visual Analogue Scale

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Cancer Center, Taipei County, Taiwan